CLINICAL TRIAL: NCT05357092
Title: Evaluation of Presurgical Orthopedics in Patients With Cleft Lip and/or Palate, a Randomized Controlled Clinial Trial.
Brief Title: Effects of AlignBabyCleft (ABaCleft)
Acronym: (ABaCleft)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The 360º Cleft Project -ABa
Record Dates: First submitted 2022-03-22; First posted 2022-05-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-11

CONDITIONS: Cleft Lip; Cleft Palate
Keywords: "cleft lip"; " Cleft palate"; "presurgical orthopedics"
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Patients treated with clear aligners to bring cleft segments closer previous to primary lip surgery.
  An average of 15 aligners will be needed although it depends on the cleft.
  Interventions: Device: Appliance. Orthodontic appliance to carry out dentoalveolar movement
- Gold Standard (No Intervention): The reference therapeutic action (no pre-surgical orthopedic intervention previous to primary lip surgery)

INTERVENTIONS:
Device: Appliance. Orthodontic appliance to carry out dentoalveolar movement — A digital 3D model obtained with a 3D scanner: (T1,baseline), (T2, aprox 8 weeks), and at the end of othopedic treatment previous to primary lip surgery (T3, aprox 16 weeks).
  Once a week, clinical check.
  Other Names: Clear Aligners
  Arms: Intervention group

SUMMARY:
Since the appearance of presurgical infant orthopedic (PSIO) as a treatment for patients with cleft lip and palate ( CLP) , numerous techniques have been described with the aim of aligning the displaced alveolar segments and restoring the position of the lateral cartilage, thus improving the results of primary surgery. Currently, the most used technique in the different protocols is the nasoalveolar molding (NAM) described by Grayson, from which variants and modifications have emerged in order to improve its results and provide greater comfort for both the patient and their caregivers.

However, the main drawback of traditional acrylic NAM is the need for sequential addition of acrylic to reduce the size of the indentation. These weekly adjustments consume time and resources for the caregiver and the orthodontist. Likewise, it has been observed that acrylic resin can cause inflammation, irritation and gingival ulceration due to excessive pressure.

PSIO treatment in newborns is a complex procedure that could benefit from simplification through digitization, providing accuracy and precision, avoiding risks such as respiratory obstruction and cyanosis that can be produced by taking impressions with alginates or silicones, most of them needing to be performed under general anesthesia.

Until now, infant care has been left out of such digitization, despite the fact that the majority of babies who need early orthodontic treatment often suffer from craniofacial disorders. However, in recent years numerous advances have been made in this type of treatment, both in taking records, and in the application of more physiological, lighter and constant forces, providing greater comfort, better acceptance and less pain for the patient . These changes represent a great advance applicable to patients with CLP.

DETAILED DESCRIPTION:
The AlingBabyCleft (AbaCleft) trial will be designed as a randomized controlled clinical trial, with an investigator blinded, superiority trial with two parallel arms.

Active treatment will be planned as soon as possible after the patient's birth, once the patient has been diagnosed with CLP and once the caregivers have been duly informed about the clinical trial, as well as its advantages and disadvantages.

The main objective (MO) of this study is to analyze the changes that occur in the dental arches of a newborn patient, diagnosed with CLP, with PSIO performed with transparent aligners, a technique that is very different from that performed in this type of surgery in patients to date.

ELIGIBILITY:
Inclusion Criteria:

Patients selected for the clinical trial must meet these criteria after randomization:

* All patients born at term, without any syndrome associated with CLP, aged between 7 days and one month of life, referred from the different hospitals of the Spanish Health System, will be included in the study.
* No distinction will be made on the basis of race or ethnic group to which the participants belong.
* Any patient will be discriminated due to distance from their place of residence.
* Participants must agree to attend regular check-ups.
* All patients who agree to be part of the experimental study must previously sign the specific informed consent designed for this purpose.

Exclusion Criteria:

* Caregivers who are not fluent in the Spanish language will be excluded in order to understand and assimilate all the instructions provided for treatment compliance.
* Patients who do not comply with the regimen of visits to the orthodontic department, and for whom a correct control of the evolution of the treatment cannot be guaranteed, will be excluded from the study.
* Lack of collaboration or non-compliance with the use of the clear aligners will also be considered grounds for exclusion.
* Patients with soft tissue bands should also be excluded from our study.

Ages: 7 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-11-21 (Estimated); Primary Completion 2027-11-21 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Inter arch dimensions | 1 year ( Primary completion)
  For the analysis of inter-arch dimensions and their clinical significance, 15 arch analysis variables will be studied.
  An intraoral scan of the patient will be performed to obtain the digitized models in different phases of the treatment. Before the start of treatment with PSIO (0 months), before lip closure (3 months), before palate closure surgery (6 months).
  The following variables will be recorded anonymously for each patient:
  * Measurements of arch width: Transverse dimension ( measured in millimeters).
  * Measurementes of arch depth: Sagital dimension ( mesaured in millimeters).
  * Alveolar arch length (measured in millimeters).
  * Arch circumference ( measured in millimeters).
  * Measurements of alignment of the segments ( measured in millimeters).

SECONDARY OUTCOMES:
Positive aspects for caregivers | 1 year ( primary completion)
  Surveys of caregivers reflecting, for later analysis, certain aspects considered positive, provided by the treatment and which will be evaluated as variables in the study.
  For the answers, a scale with 4 points will be used:
  1. Very satisfactory, very happy, more than adequate.
  2. Satisfactory, happy, adequate.
  3. Unsatisfactory, unhappy, inadequate.
  4. Very unsatisfactory, very unhappy, very inadequate.

CONTACTS AND LOCATIONS:
Overall Officials: ROSA YAÑEZ VICO, Study Director — COMPLUTENSE UNIVERITY OF MADRID

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allareddy V, Shusterman S, Ross E, Palermo V, Ricalde P. Dentofacial Orthopedics for the Cleft Patient: The Latham Approach. Oral Maxillofac Surg Clin North Am. 2020 May;32(2):187-196. doi: 10.1016/j.coms.2020.01.002. Epub 2020 Feb 17. PMID 32081579
- [Result] Ball JV, DiBiase DD, Sommerlad BC. Transverse maxillary arch changes with the use of preoperative orthopedics in unilateral cleft palate infants. Cleft Palate Craniofac J. 1995 Nov;32(6):483-8. doi: 10.1597/1545-1569_1995_032_0483_tmacwt_2.3.co_2. PMID 8547288
- [Result] Berkowitz S, Mejia M, Bystrik A. A comparison of the effects of the Latham-Millard procedure with those of a conservative treatment approach for dental occlusion and facial aesthetics in unilateral and bilateral complete cleft lip and palate: part I. Dental occlusion. Plast Reconstr Surg. 2004 Jan;113(1):1-18. doi: 10.1097/01.PRS.0000096710.08123.93. PMID 14707617
- [Result] Fuchigami T, Kimura N, Kibe T, Tezuka M, Amir MS, Suga H, Takemoto Y, Hashiguchi M, Maeda-Iino A, Nakamura N. Effects of pre-surgical nasoalveolar moulding on maxillary arch and nasal form in unilateral cleft lip and palate before lip surgery. Orthod Craniofac Res. 2017 Nov;20(4):209-215. doi: 10.1111/ocr.12199. Epub 2017 Sep 18. PMID 28921849
- [Result] Adali N, Mars M, Petrie A, Noar J, Sommerlad B. Presurgical orthopedics has no effect on archform in unilateral cleft lip and palate. Cleft Palate Craniofac J. 2012 Jan;49(1):5-13. doi: 10.1597/11-030. Epub 2011 Aug 8. PMID 21823827
- [Result] Mars M, Asher-McDade C, Brattstrom V, Dahl E, McWilliam J, Molsted K, Plint DA, Prahl-Andersen B, Semb G, Shaw WC, et al. A six-center international study of treatment outcome in patients with clefts of the lip and palate: Part 3. Dental arch relationships. Cleft Palate Craniofac J. 1992 Sep;29(5):405-8. doi: 10.1597/1545-1569_1992_029_0405_asciso_2.3.co_2. PMID 1472517
- [Result] Prahl C, Prahl-Andersen B, Van't Hof MA, Kuijpers-Jagtman AM. Presurgical orthopedics and satisfaction in motherhood: a randomized clinical trial (Dutchcleft). Cleft Palate Craniofac J. 2008 May;45(3):284-8. doi: 10.1597/07-045.1. PMID 18452361
- [Result] Al Khateeb KA, Fotouh MA, Abdelsayed F, Fahim F. Short-Term Efficacy of Presurgical Vacuum Formed Nasoalveolar Molding Aligners on Nose, Lip, and Maxillary Arch Morphology in Infants With Unilateral Cleft Lip and Palate: A Prospective Clinical Trial. Cleft Palate Craniofac J. 2021 Jul;58(7):815-823. doi: 10.1177/1055665620966189. Epub 2020 Oct 27. PMID 33107321
- [Result] Gong X, Dang R, Xu T, Yu Q, Zheng J. Full Digital Workflow of Nasoalveolar Molding Treatment in Infants With Cleft Lip and Palate. J Craniofac Surg. 2020 Mar/Apr;31(2):367-371. doi: 10.1097/SCS.0000000000006258. PMID 32049908
- [Result] Batra P, Gribel BF, Abhinav BA, Arora A, Raghavan S. OrthoAligner "NAM": A Case Series of Presurgical Infant Orthopedics (PSIO) Using Clear Aligners. Cleft Palate Craniofac J. 2020 May;57(5):646-655. doi: 10.1177/1055665619889807. Epub 2019 Dec 4. PMID 31795731